CLINICAL TRIAL: NCT00342381
Title: Fatigue in Multiple Sclerosis: Evaluated With 3 Tesla MRI and Transcranial Magnetic Stimulation
Brief Title: Fatigue in Multiple Sclerosis: Evaluated With 3 MRI and Transcranial Magnetic Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Multiple Sclerosis Society (Unknown)
Responsible Party: Henning Andersen, Dep of neurology, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20060003
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Motor fatigue; Cognitive fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Amifampridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3.4 diaminopyridine (Active Comparator): Single dose 3,4 diaminopyridine
  Interventions: Drug: 3,4-diaminopyridine
- Placebo (Placebo Comparator): Two tablets identical to active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3,4-diaminopyridine — Single dose 3,4 diaminopyridine
  Arms: 3.4 diaminopyridine
Drug: Placebo — Single dose placebo treatment
  Other Names: n/d
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate fatigue in patients with multiple sclerosis (MS) and to determine the correlation between the symptom and cerebral changes.

DETAILED DESCRIPTION:
Only recruiting from:

Department of Neurology, Aarhus University Hospital, Denmark

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting-multiple sclerosis (RR-MS) according to Poser criteria
* EDSS: max 3.5
* Right handed
* Normal function of the right hand

Exclusion Criteria:

* Disease interfering with MS
* Known dementia
* Drug or alcohol abuse
* Treatment with psychoactive drugs within one week before study entry
* Major changes of medical treatment within 3 weeks before study entry
* Attack within 4 weeks before study entry
* Pregnancy
* Conditions interfering with 3,4-diaminopyridine treatment
* Conditions interfering with MRI
* Conditions interfering with transcranial magnetic stimulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Subjective fatigue (FSS) | Weeks
Maximal voluntary isometric contraction, central activation before and after exercise | at the time of investigation
Digit Symbol-Coding scores | Weeks
Changes in normal appearing white matter and normal appearing gray matter (MRS-, MTI- and DTI- parameters) | at the time of MRI
Cortical atrophy | at the time of MRI
Intracortical inhibition/facilitation determined by transcranial magnetic stimulation (+/- 3,4-diaminopyridine) | at the time of investigation

SECONDARY OUTCOMES:
Subjective fatigue (MFI-20, Danish version) | Weeks
Rapid voluntary twitches | at the time of investigation
6 minute walk test | at the time of investigation
9-hole peg test | at the time of investigation
WAIS/WMS tests | at the time of investigation
WHO-5 Questionnaire | at the time of investigation
Major Depression Inventory | at the time of investigation
Lesion load | at the time of MRI
Whole brain atrophy | at the time of MRI
Subjective fatigue (VAS) | at the time of investigation

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, DMSc, Principal Investigator — Aarhus University Hospital; Johannes Jacobsen, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Neurology, Aarhus, Denmark